CLINICAL TRIAL: NCT04934280
Title: Diagnostic Yield of Transvaginal Ultrasonography Versus Sonohysterography in the Evaluation of Ceserean Section Niche.
Brief Title: Diagnostic Yield of Transvaginal Ultrasonography Versus Sonohysterography in Detection of Ceserean Section Niche
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Radwa Ahmed Elbahy Mohamed, Resident at diagnostic radiology department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-06-10
Record Dates: First submitted 2021-06-16; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cesarean Section Niche Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2D transvaginal ultrasonography (Other)
  Interventions: Diagnostic Test: sonohysterography

INTERVENTIONS:
Diagnostic Test: sonohysterography — saline infusion transvaginally followed by 2D transvaginal ultrasound imaging

SUMMARY:
The aim of this study is to compare the identification of CS scar niche between 2D transvaginal ultrasonography alone and with the use of saline infusion as a contrast. Does it differ in the measurements and identification or not.

DETAILED DESCRIPTION:
Cesarean section (CS) rate is increasing in recent practice with a corresponding increase in associated complication. One of these complications is the CS scar defect or 'niche'. A niche forms after CS at the site of hysterotomy of the anterior uterine wall. Recently, it has been demonstrated that niche may be the causative factor for abnormal uterine bleeding, dysmenorrhea, obstetric complications in subsequent pregnancies and possibly subfertility. Therefore, the accurate measurement and description of a niche is becoming increasingly important, for the clinical assessment of gynecological symptoms and for the planning of possible surgical treatment.A niche can be examined using two- (2D) or three- (3D) dimensional transvaginal sonography (TVS), with or without saline or gel contrast, magnetic resonance imaging and hysteroscopy. We will examine about 30 patients of non pregnant women with previous CS having gynecological complications or seeking fertility. All participants will be subjected to 2D vaginal examination to exclude uterine pathology followed by 2D transvaginal ultrasonography with saline infusion using 10-20 ml of sterile Na Cl 0.9% solution injected through the cervix using a 2 mm sterile disposable catheter or IOL Foley catheter. The procedure will be done postmenstrually.

ELIGIBILITY:
Inclusion Criteria:

* women with previous CS section scar seeking pregnancy or having gynecological complications

Exclusion Criteria:

* women having other gynecological pathology other than niche

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
accurate evaluation of CS section niche | 6 months from the date of approval
  comparison of imaging CS niche by 2D transvaginal US and sonohysterography

IPD SHARING:
Plan to Share IPD: No